CLINICAL TRIAL: NCT04645472
Title: Accurate Positioning of CT-Ultrasound Fusion in PCNL Puncture Guidance
Brief Title: CT-Ultrasound Fusion in Guiding PCNL Puncture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhenyu Wu (Other)
Responsible Party: Sponsor-Investigator, Zhenyu Wu, Medical Doctor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: 2020-KY-021
Record Dates: First submitted 2020-11-25; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT-Ultrasound group
  Interventions: Device: CT-Ultrasound

INTERVENTIONS:
Device: CT-Ultrasound — For patients with kidney stones who are planning to undergo PCNL, perform a preoperative simulated CT-ultrasound fusion examination to further clarify the condition of the kidney stones and simulate and optimize the puncture route. Apply CT- Ultrasound fusion precise positioning to guide the intraoperative PCNL puncture process.

SUMMARY:
Kidney stone is a common urological disease. Percutaneous nephrolithotomy (PCNL) is an important method for the treatment of kidney stones. The accuracy of puncture positioning affects the PCNL stone free rate and intraoperative/postoperative complications. Currently, PCNL puncture positioning methods are mainly X-ray-guided or ultrasound-guided. The main disadvantage of X-ray is the lack of soft tissue imaging, and the problem of low puncture accuracy. Although ultrasound is a commonly used real-time imaging tool, the image is not intuitive enough, and the puncture path is deviated from actual requirements . In order to improve the accuracy of PCNL puncture, this study intends to import CT images of both kidneys into a novel ultrasound machine through an image fusion system to achieve CT-ultrasound image fusion, and to simulate the puncture route to guide the PCNL puncture process. The study is mainly divided into two parts: (1) For patients with kidney stones who are planning to undergo PCNL, perform a preoperative simulated CT-ultrasound fusion examination to further clarify the condition of the kidney stones and simulate and optimize the puncture route; (2) Apply CT- Ultrasound fusion precise positioning to guide the intraoperative PCNL puncture process. On the basis of traditional ultrasound images, the CT-ultrasound fusion image display is added to provide the optimal puncture route to explore the effectiveness and safety of CT-ultrasound fusion precise positioning in PCNL puncture.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years old, gender is not limited, and can tolerate surgery; (2) Kidney stone patients who intend to undergo PCNL surgery; (3) Have kidney CT data; (4) Volunteer to participate and sign informed consent.

Exclusion Criteria:

* (1) Uncontrollable systemic hemorrhagic disease; (2) Severe spinal deformity, severe hip deformity, and difficult lithotomy position; (3) Uncontrolled urinary tract infection; (4) Cavity caused by any urinary system anatomy Internal surgery cannot be performed; (5) Pregnant women, women who plan to become pregnant within 3 months, and lactating women; (6) Patients with severe heart, lung and brain diseases that cannot tolerate surgery; (7) The investigator judges that the patient is not suitable for participating in this study , Including (but not limited to): known to be carrying human immunodeficiency virus or suffering from AIDS; suffering from mental illness; infectious diseases, etc.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We plan to enroll 50 patients to explore the effectiveness and safety of CT-ultrasound fusion in guiding PCNL puncture positioning.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | in a week
  Stone free rate in a week

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenyu Wu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizvi SAH, Hussain M, Askari SH, Hashmi A, Lal M, Zafar MN. Surgical outcomes of percutaneous nephrolithotomy in 3402 patients and results of stone analysis in 1559 patients. BJU Int. 2017 Nov;120(5):702-709. doi: 10.1111/bju.13848. Epub 2017 Apr 17. PMID 28303631
- [Background] Kalogeropoulou C, Kallidonis P, Liatsikos EN. Imaging in percutaneous nephrolithotomy. J Endourol. 2009 Oct;23(10):1571-7. doi: 10.1089/end.2009.1521. PMID 19630501
- [Background] Ghani KR, Andonian S, Bultitude M, Desai M, Giusti G, Okhunov Z, Preminger GM, de la Rosette J. Percutaneous Nephrolithotomy: Update, Trends, and Future Directions. Eur Urol. 2016 Aug;70(2):382-96. doi: 10.1016/j.eururo.2016.01.047. Epub 2016 Feb 11. PMID 26876328
- [Background] Xu ZF, Xie XY, Kuang M, Liu GJ, Chen LD, Zheng YL, Lu MD. Percutaneous radiofrequency ablation of malignant liver tumors with ultrasound and CT fusion imaging guidance. J Clin Ultrasound. 2014 Jul-Aug;42(6):321-30. doi: 10.1002/jcu.22141. Epub 2014 Feb 25. PMID 24615771
- [Background] Da Rosa MR, Milot L, Sugar L, Vesprini D, Chung H, Loblaw A, Pond GR, Klotz L, Haider MA. A prospective comparison of MRI-US fused targeted biopsy versus systematic ultrasound-guided biopsy for detecting clinically significant prostate cancer in patients on active surveillance. J Magn Reson Imaging. 2015 Jan;41(1):220-5. doi: 10.1002/jmri.24710. Epub 2014 Jul 21. PMID 25044935